CLINICAL TRIAL: NCT01776177
Title: A REAL-LIFE RETROSPECTIVE ANALYSIS OF CLINICAL CHARACTERISTICS AND IMPACT OF LONG-TERM TREATMENT WITH OMALIZUMAB WITH EMPHASIS ON MARKERS OF RESPONSE IN A CLINICAL PRACTICE IN APPROXIMATELY 240 PATIENTS WITH MODERATE-TO-SEVERE ALLERGIC ASTHMA
Brief Title: The REALITY Study - a Real-life Long-term Analysis of Xolair Therapy
Acronym: The Reality
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Joseph D. Diaz, MD (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph D. Diaz, MD, Medical Director, Allergy & Asthma Research Center, San Antonio, TX
Organization: Allergy & Asthma Research Center, San Antonio, TX (Industry)
Other Study IDs: ML28357
Record Dates: First submitted 2012-09-18; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Allergic Asthma
Keywords: Allergic asthma; Omalizumab therapy; IgE profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continue Therapy Group: Patients who continued to recieve Omalizumab therapy beyond 6 month period
- Discontinued Therapy group: Patients who discontinued Omalizumab therapy prior to 6 month period from the start of therapy

SUMMARY:
The primary objective is to assess the clinical effectiveness of long-term omalizumab therapy in 240 patients treated over an 8 year period in a real-life clinical setting and to compare the pre- and post-treatment clinical characteristics to identify and better understand the markers of response to omalizumab.

To date, there are no established criteria for identifying 'response' to omalizumab therapy. Currently, the commonly accepted clinical criterion for omalizumab treatment response is the physician's overall assessment, GETE (Global Evaluation of Treatment Effectiveness). Most clinical trials have evaluated the efficacy of omalizumab treatment after a 16 week treatment period and lack the impact of long-term omalizumab therapy.

Investigators propose multiple approach modules to better assess and identify 'response' and to define 'responders' to omalizumab and evaluate the long-term impact in a real-world clinical practice. Besides evaluating individual outcome variables, it is important to attempt the 'clustering of variables' to further investigate if any baseline clinical phenotypes are predictive of better response enabling us to refine the patient population who will gain most benefit from therapy.

DETAILED DESCRIPTION:
Medical records from 240 omalizumab-treated patients will be evaluated. Comprehensive data will be collected for any asthma-related event (see evaluation criteria below), omalizumab dose, asthma-medications, spirometry, asthma control test (ACT) and any respiratory infection and/or antibiotic use since last visit. Data will be analyzed to compare the clinical phenotypes and outcome among patients to identify, characterize and define 'responders' and 'non-responders' to omalizumab. Periodic assessments for demonstrated level of response and need for continued therapy will be evaluated quarterly. Also, real-life patient adherence data to long-term omalizumab therapy will be analyzed and the factors for withdrawal and non-adherence will be identified.

Reduction in annualized rate of asthma exacerbation, steroid bursts and oral steroid dosage, ER/unscheduled doctor's visits, hospitalization and improvement in spirometry and ACT score and review of asthma medications will be evaluated quarterly. 'Cluster analysis' will be performed by grouping variables (such as age, asthma duration and severity, dosage, therapy duration, sensitization profile, IgE levels etc.) in effort to identify groups of responders.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-to-severe persistent allergic asthmatic patients with inadequate asthma control
2. Received Omalizumab therapy per steps 5 & 6 of the NHLBI guidelines
3. Positive skin test or in-vitro specific IgE to perennial allergens
4. Measured baseline total serum IgE level (within 1 year from first dose)
5. Patient followed at AAIAST/AARC (from February 2004 to December 2011)

Exclusion Criteria:

* N/A; retrospective study

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single-center, retrospective study; total 240 patients. All 240 patients with moderate-to-severe allergic asthma who have received Omalizumab therapy at AAIAST/AARC [from February 2004 to December 2011].
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Integrated Asthma control assessment(Change From Baseline) | February 2004 to December 2011. [ Time Frame: Baseline, 3-, 6-, 9-, 12-, 18-, 24-, 36-, 48-, 60-, 72- months of therapy]
  Data from 240 omalizumab-treated patients will be collected for for the above stated time frame for pre- and post-treatment periods. The parameters assessed will be for Spirometry, Asthma Medications, ACT score.
Integrated Asthma severity assessment (Change From Baseline): [ Time Frame: Baseline, 3-, 6-, 9-, 12-, 18-, 24-, 36-, 48-, 60-, 72- months of therapy] | February 2004 to December 2011. [ Time Frame: Baseline, 3-, 6-, 9-, 12-, 18-, 24-, 36-, 48-, 60-, 72- months of therapy]
  Data from 240 omalizumab-treated patients will be collected for for the above stated time frame for pre- and post-treatment periods. The parameters assessed will be for Asthma exacerbation, Steroid bursts, Oral steroid, Hospitalization/ ER visits.

SECONDARY OUTCOMES:
'Clustering' of outcome variables | February 2004 to December 2011. The time frame of all subjects is variable ranging from 3 months to 8 years depending on the duration the patients were on omalizumab therapy.
  Data from 240 omalizumab-treated patients will be collected for the 'secondary outcome measure' parameters (as stated above).
  1. Age
  2. Asthma duration and severity
  3. Therapy duration
  4. Drug dosage
  5. IgE levels Data will be analyzed to compare the clinical phenotypes and outcome among patients to identify, characterize and define 'responders' and 'non-responders' to omalizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Diaz, MD, Principal Investigator — Allergy & Asthma Research Center, San Antonio, TX
Locations (1):
- Allergy & Asthma Research Center (AARC), San Antonio, Texas, United States

REFERENCES:
- [Derived] Singh H, Peters JI, Kaur Y, Maselli DJ, Diaz JD. Long-term evaluation of response to omalizumab therapy in real life by a novel multimodular approach: The Real-life Effectiveness of Omalizumab Therapy (REALITY) study. Ann Allergy Asthma Immunol. 2019 Nov;123(5):476-482.e1. doi: 10.1016/j.anai.2019.07.026. Epub 2019 Aug 2. PMID 31382020